CLINICAL TRIAL: NCT06750263
Title: Effects of Balance Exercises With and Without Clamshell Exercises on Physical Performanace and Balance After Menopause
Brief Title: Effects of Balance Exercises With and Without Clamshell Exercises After Menopause
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0521
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Menopause
Keywords: Balance; Clamshell; Postmenupause

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance exercises with clamshell (Experimental): balance was assessed by the Berg's Balance Scale exercise. Participants were instructed to walk (step) from one end of the mat to the other according to the step pattern provided. When reached the end of the mat, instructed to return to their starting position by walking normally off the mat and starting the next stepping. repeat every sequence five times and then started a new pattern. Duration would be 30 min. clamshell exercises a Participants were instructed to lie on their side with the weaker limb facing upwards. Both hips were flexed at 45 degrees, knees flexed at 90 degrees, and neither the feet nor the back were in contact with the wall. While keeping both heels and the first metatarsal head together, participants were instructed to separate their knees and rotate the weaker limb upward. They were advised not to tilt the limb backwards and to maintain a neutral pelvic position 3,5 sets for 10 repetations twice a week for 12 weeks
  Interventions: Other: Balance exercise with clamshell; Other: Balance exercise
- balance exercise (Active Comparator): Group B will be recieve balance exercises balance was assessed by the Berg's Balance Scale exercise include square stepping exercises The SSE comprised a progression of forward, in reverse, sidelong, and inclining steps. Participants were instructed to walk (step) from one end of the mat to the other according to the step pattern provided. When they reached the end of the mat, they were instructed to return to their starting position by walking normally off the mat and starting the next stepping. Each participant repeated every sequence five times and then started a new pattern. Duration of exercise would be 30 min
  Interventions: Other: Balance exercise

INTERVENTIONS:
Other: Balance exercise with clamshell — balance was assessed by the Berg's Balance Scale exercise. Participants were instructed to walk (step) from one end of the mat to the other according to the step pattern provided. When reached the end of the mat, instructed to return to their starting position by walking normally off the mat and starting the next stepping. repeat every sequence five times and then started a new pattern. Duration would be 30 min. clamshell exercises a Participants were instructed to lie on their side with the weaker limb facing upwards. Both hips were flexed at 45 degrees, knees flexed at 90 degrees, and neither the feet nor the back were in contact with the wall. While keeping both heels and the first metatarsal head together, participants were instructed to separate their knees and rotate the weaker limb upward. They were advised not to tilt the limb backwards and to maintain a neutral pelvic position 3,5 sets for 10 repetations twice a week for 12 weeks
  Arms: Balance exercises with clamshell
Other: Balance exercise — Participants were instructed to lie on their side with the weaker limb facing upwards. Both hips were flexed at 45 degrees, the knees were flexed at 90 degrees, and neither the feet nor the back were in contact with the wall. While keeping both heels and the first metatarsal head together, participants were instructed to separate their knees and rotate the weaker limb upward. They were advised not to tilt the limb backwards and to maintain a neutral pelvic position 3,5 sets for 10 repetations twice a week for 12 weeks

SUMMARY:
Exercise-based balance intervention is structured program of physical exercises intended to enhance balance, stability, and clamshell exercises are known as an exercise-based balance intervention. A crucial component of physical therapy and fitness regimens targeted at enhancing stability, reducing the risk of falls, and promoting general physical health is exercise-based balance therapies. Women's ability to function both physically and mentally can be significantly impacted by menopause. To find out the effects of an exercise based balance intervention on physical and clamshell exercises after menopause Certain consequences can be lessened by address these alterations with focused interventions.These will be a randomized clinical trial and will be conducted in Bhawalpur Victoria Hospital and Mehran Rehab Clinic. This study will be completed in the time duration of 10 months after the approval of Synopsis. Non probability convenience sampling technique will be used and participants will be recruited in study after the randomization.80 participants with age between 50-65 years will be included in the study according to the inclusion criteria. Group A will receive balance exercises and clamshell exercises Group B will be recieve only balance exercises the tool that will be used are the sit and raised test , y balance test, Romberg test for check the balance. Timed raised chair task for check the strength . timed up and go for check the mobility . heel shin touch test for check the coordination. Time shuttle runs for check the speed. Step test for check the power after data collection, data will be analyzed by using SPPSS 26.

ELIGIBILITY:
Inclusion Criteria:

* age 65 years or older;
* having significant concerns about their balance
* participants to be living independently in the community
* Berg's Balance Scale scores more than 41/56 indicating minimal fall risk were included in the study

Exclusion Criteria:

* Participants were excluded from the study if their vision was compromised so that they were unable to see objects on the floor or recognize the instructor's movements

  * progressive neurologic disease which could impair balance
  * hypertensive
* unable to understand, speak, or hear

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Time shuttle run | baseline and fourth week
  A maximal multistage 20 m shuttle run test was designed to determine the maximal aerobic power of menopausal females Subjects run back and forth on a 20 m course and must touch the 20 m line; at the same time The reliability of the interval shuttle run test (ISRT) as a submaximal and maximal field test to measure intermittent endurance capacity was examined. ISRT. Relative reliability was high (intraclass correlation coefficient ≥ 0.86). A maximal multistage 20 m shuttle run test was designed to determine the maximal aerobic power of menopausal females Subjects run back and forth on a 20 m course and must touch the 20 m line; at the same time. The reliability of the interval shuttle run test (ISRT) as a submaximal and maximal field test to measure intermittent endurance capacity was examined. ISRT.
Time up and go | baseline and fourth week
  TUG measures the time a person needs to get up out of a chair, walk three meters and return to the chair. This is measured in seconds with a handheld stopwatch. Patients performed the TUG two times and for each patient, the mean of the two time measurements would be a score of less than or equal to 20 seconds on the TUG was considered a normal score

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Riphah International University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh GS, Delextrat A, Bibbey A. The comparative effect of exercise interventions on balance in perimenopausal and early postmenopausal women: A systematic review and network meta-analysis of randomised, controlled trials. Maturitas. 2023 Sep;175:107790. doi: 10.1016/j.maturitas.2023.107790. Epub 2023 Jun 16. PMID 37343343
- [Background] Shojaa M, Von Stengel S, Schoene D, Kohl M, Barone G, Bragonzoni L, Dallolio L, Marini S, Murphy MH, Stephenson A, Manty M, Julin M, Risto T, Kemmler W. Effect of Exercise Training on Bone Mineral Density in Post-menopausal Women: A Systematic Review and Meta-Analysis of Intervention Studies. Front Physiol. 2020 Jun 23;11:652. doi: 10.3389/fphys.2020.00652. eCollection 2020. PMID 32655410
- [Background] Shubert TE, McCulloch K, Hartman M, Giuliani CA. The effect of an exercise-based balance intervention on physical and cognitive performance for older adults: a pilot study. J Geriatr Phys Ther. 2010 Oct-Dec;33(4):157-64. PMID 21717919